CLINICAL TRIAL: NCT02685852
Title: A Pilot Study Evaluating Exenatide for the Treatment of Postprandial Hyperinsulinemic Hypoglycemia Post-RYGB
Brief Title: Evaluating Exenatide for the Treatment of Postprandial Hyperinsulinemic Hypoglycemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1503M65841
Record Dates: First submitted 2016-01-19; First posted 2016-02-19 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Hyperinsulinemic Hypoglycemia
MeSH Terms: conditions — Congenital Hyperinsulinism | interventions — Exenatide; Acarbose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Exenatide (5mcg) + Acarbose Placebo (Active Comparator): Exenatide (5 mcg) 30 minutes before the high-carb meal is delivered and acarbose placebo immediately prior to the high-carb meal
  Interventions: Drug: Exenatide; Drug: Acarbose Placebo
- Arm 2: Exenatide (5mcg) + Acarbose (25mg) (Active Comparator): Exenatide (5 mcg) 30 minutes before the high-carb meal is delivered and acarbose (25 mg) immediately prior to the high-carb meal
  Interventions: Drug: Exenatide; Drug: Acarbose
- Arm 3: Exenatide Placebo + Acarbose (25mg) (Placebo Comparator): Exenatide placebo 30 minutes before the high-carb meal is delivered and acarbose (25 mg) immediately prior to the high-carb meal
  Interventions: Drug: Acarbose; Drug: Exenatide Placebo

INTERVENTIONS:
Drug: Exenatide — Exenatide at a dose of 5 mcg
  Other Names: Byetta
  Arms: Arm 1: Exenatide (5mcg) + Acarbose Placebo; Arm 2: Exenatide (5mcg) + Acarbose (25mg)
Drug: Acarbose — Acarbose at a dose of 25 mg
  Arms: Arm 2: Exenatide (5mcg) + Acarbose (25mg); Arm 3: Exenatide Placebo + Acarbose (25mg)
Drug: Exenatide Placebo — Placebo for Exenatide
  Arms: Arm 3: Exenatide Placebo + Acarbose (25mg)
Drug: Acarbose Placebo — Placebo for Acarbose
  Arms: Arm 1: Exenatide (5mcg) + Acarbose Placebo

SUMMARY:
The purpose of the study is to evaluate the effectiveness of exenatide in adults experiencing episodes of hyperinsulinemic hypoglycemia following Roux-en-Y bariatric surgery.

DETAILED DESCRIPTION:
Roux-en-Y gastric bypass surgery (RYGB) is one of the most common bariatric surgeries in the United States and is generally highly effective for weight loss. Unfortunately, among the potential complications is hyperinsulinemic hypoglycemia. Though the prevalence of this disorder has not been fully characterized, it can be associated with debilitating symptoms which severely impact quality of life and can be life-threatening. The underlying pathophysiology of hyperinsulinemic hypoglycemia likely involves a mismatch in the amount of insulin secreted in response to mealtime carbohydrate absorption. It has been observed that the ingestion of a high carbohydrate load often leads to a modest rise in post-prandial glucose levels followed by an inappropriately exaggerated insulin release among individuals with this condition. Low carbohydrate diet sometimes provides full or partial relief of the symptoms.

Standard medical management for RYGB associated postprandial hyperinsulinemic hypoglycemia includes acarbose, which partially reduces carbohydrate absorption from the gut, and diazoxide, which directly inhibits insulin release from pancreatic beta cells. However, the medical options are not reliably effective, leading some individuals to reverse RYGB, which also may not be effective, or even undergo partial pancreatectomy, risking additional complications such as diabetes. Much more reliably effective treatments are needed for this special population who develop this bariatric surgical complication.

Potential mechanisms contributing to the mismatched insulin secretion post RYGB include decreased systemic and adipose tissue inflammation, and increased insulin receptor expression in liver and skeletal muscle, and increases in adiponectin.

ELIGIBILITY:
Inclusion Criteria:

1. must have undergone RYGB and subsequently developed post-prandial hypoglycemia (defined as at least 3 episodes over a six-month period with documented capillary blood sugars [<60 mg/dL with hypoglycemic symptoms). Subjects may also have had a formal mixed meal tolerance test with post meal blood sugar <60 mg/dL.
2. Subjects who otherwise meet the study criteria above with hypoglycemia symptoms but who do not have documented hypoglycemia by plasma measurement may undergo a screening visit to document the requisite levels for consideration into the study.

Exclusion Criteria:

1. Chronic or acute diseases of the liver.
2. Chronic or acute diseases of the pancreas (including type 1 diabetes or pancreatitis or a history of pancreatitis). Subjects may have a diagnosis of type 2 diabetes but must no longer require diabetes medication.
3. Chronic or acute diseases of the kidneys.
4. Known malignancies and must not have a family history of medullary thyroid cancer.
5. History of pre-RYGB hypoglycemia symptoms or low documented plasma glucose preoperatively.
6. Pregnant or plans to become pregnant throughout study duration
7. Breastfeeding
8. Medication exclusions in addition to the current use of diabetes medications. Subjects will be excluded if they have previously taken GLP-1 agonists.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-02; Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Glucose area under the curve (AUC) following treatment for each 4-hour test period | During the 4-hour test period
  Each time point (15, 30, 45, 60, 90, 120, 180 and 240 minutes) will be used to calculate AUC using the trapezoidal method.
Presence of hypoglycemia | 15, 30, 45, 60, 90, 120, 180 and 240 minutes
  If at each time-point (15, 30, 45, 60, 90, 120, 180 and 240 minutes) plasma glucose is <60 mg/dL, participants will be defined as hypoglycemic

SECONDARY OUTCOMES:
Minimum post-prandial blood sugar level (mg/dL) | post meal test
  The lowest post-prandial blood glucose level at any time point (15, 30, 45, 60, 90, 120, 180 and 240 minutes) may be used as the minimum post-prandial blood sugar level (mg/dL).
Change in post-prandial blood glucose from 0min to 120min | 0min to 120min
  % change in blood glucose 0min to 120min
Change in post-prandial Insulin levels (mcg/mL) | 0min to 120min
  % change in insulin 0min to 120min

CONTACTS AND LOCATIONS:
Overall Officials: Shalamar D Sibley, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States